CLINICAL TRIAL: NCT05447039
Title: Value of Montelukast as a Potential Treatment of Post COVID-19 Persistent Cough: A Randomized Controlled Pilot Study
Brief Title: Value of Montelukast as a Potential Treatment of Post COVID-19 Persistent Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AssiutU21-1
Record Dates: First submitted 2022-07-03; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Post COVID-19
Keywords: Montelukast; cough; cough severity
MeSH Terms: conditions — Cough | interventions — montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Montelukast treated (Active Comparator)
  Interventions: Drug: Montelukast Sodium Tablets
- Standard treatment (No Intervention)

INTERVENTIONS:
Drug: Montelukast Sodium Tablets — intervention group received standard cough therapy+ Montelukast 10 mg/day for 14 days
  Other Names: Montelukast
  Arms: Montelukast treated

SUMMARY:
As of September 2020, the COVID-19 pandemic has affected millions of people in 196 countries and left hundreds of thousands dead. After recovery it was found that up to 32% of cases had 1 or 2 symptoms, 55% had 3 or more Post-COVID-19 symptoms, and persistent Post COVID-19 cough was recorded in 29.3% of cases in one study.

A recent study identified Montelukast, among the top-scoring clinically-oriented drugs likely to inhibit SARS-CoV-2 main protease. Besides its known effect that is reported to improve cough and prevent exercise-induced bronchoconstriction in asthma, many trials assessed Montelukast in the treatment of post-infectious cough and found variable effects.

Despite that the exact mechanism is not yet identified, Barré and colleagues proposed several properties of Cyst LT1 receptor antagonists that are potentially beneficial in COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Post COVID-19 persistent cough after 4 weeks of acute attack

Exclusion Criteria:

* Any contraindication to Montelukast, respiratory, cardiac disease, pregnancy, breastfeeding and use of angiotensin converting enzyme inhibitors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
cough severity index | 14 days
  Scale from mild to severe
Cough severity visual analog | 14 days
  Severity from 0-10

SECONDARY OUTCOMES:
Side effects of drug | 14 days
  Nausea, vomiting, abdominal pain, restlessness, depression

CONTACTS AND LOCATIONS:
Locations (1):
- Aliae Mohamed-Hussein, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
upon reasonable request